CLINICAL TRIAL: NCT04230681
Title: A Randomized Controlled Trial to Compare Hydromorphone vs Fentanyl in Children Undergoing Tonsillectomy Surgery
Brief Title: Hydromorphone vs Fentanyl in Children Undergoing Tonsillectomy Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201912042; UL1TR002345 (NIH)
Record Dates: First submitted 2019-12-27; First posted 2020-01-18 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea; Tonsillitis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis | interventions — Hydromorphone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl
- Hydromorphone (Active Comparator)
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Patients will be randomized to one of two opioids for the treatment of post-operative pain.
  Arms: Hydromorphone
Drug: Fentanyl — Fentanyl
  Arms: Fentanyl

SUMMARY:
A RCT to compare hydromorphone versus fentanyl for pain control following tonsillectomy or adenotonsillectomy surgery.

DETAILED DESCRIPTION:
This is a randomized clinical trial with masked assessment, comparing recovery indices for patients receiving intermediate acting versus short acting opioid analgesia using hydromorphone or fentanyl as intraoperative analgesics. An otherwise standardized anesthetic and analgesic regimen will be utilized, consistent with routine care at SLCH. Patients will be randomized 1:1 in block sizes of 5 per group. Patients will be randomized to receive either hydromorphone or fentanyl throughout the perioperative period by opening a sealed protocol envelope.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 2 to 15 years old
2. Presenting for tonsillectomy or adenotonsillectomy surgery
3. American Society of Anesthesiologists Physical Status (ASAPS) Classification 1, 2 or 3
4. Provide Informed Consent / Assent (as appropriate)

Exclusion Criteria:

1. Additional Concurrent surgeries, exclusive of myringotomy tubes, minor oral/nasal procedures (e.g. frenulectomy), and endoscopic procedures
2. Revision tonsillectomy or revision adenotonsillectomy surgery
3. Known pregnancy
4. Any condition which would make the participant, in the opinion of the investigator or the attending anesthesiologist caring for the patient, unsuitable for the study.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Montana, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman NR, Perkins JN, McNair B, Mitchell RB. Current practice patterns for sleep-disordered breathing in children. Laryngoscope. 2013 Apr;123(4):1055-8. doi: 10.1002/lary.23709. Epub 2013 Feb 4. PMID 23382017
- [Background] Brown KA. Outcome, risk, and error and the child with obstructive sleep apnea. Paediatr Anaesth. 2011 Jul;21(7):771-80. doi: 10.1111/j.1460-9592.2011.03597.x. Epub 2011 May 3. PMID 21539679
- [Background] Bhattacharyya N, Lin HW. Changes and consistencies in the epidemiology of pediatric adenotonsillar surgery, 1996-2006. Otolaryngol Head Neck Surg. 2010 Nov;143(5):680-4. doi: 10.1016/j.otohns.2010.06.918. PMID 20974339

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone; Fentanyl: Pediatric patients will be randomized to one of two arms. Arm 1 will receive intravenous hydromorphone intraoperatively following induction of general anesthesia. Arm 2 will receive intravenous fentanyl in the operating room following induction of general anesthesia.
Period: Overall Study
Arm/Group | Hydromorphone | Fentanyl
Started | 93 | 95
Completed | 90 | 90
Not Completed | 3 | 5
Not completed — Physician Decision | 2 | 3
Not completed — Investigational Pharmacy unable to provide medications in timely manner | 1 | 1
Not completed — IV inadvertently removed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Hydromorphone: Pediatric patients randomized to receive hydromorphone intravenously in the operating room.
- Fentanyl: Pediatric patients randomized to receive fentanyl intravenously in the operating room.
- Total: Total of all reporting groups
Arm/Group | Hydromorphone | Fentanyl | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 90 | 90 | 180
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 54 | 50 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 86 | 87 | 173
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 19 | 38
  White | 68 | 67 | 135
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring Rescue Intravenous Opioid
Description: Number
Time Frame: up to 6 hours post surgery
Measure: Count of Participants; unit: Participants
Groups:
- Hydromorphone: Pediatric patients randomized to hydromorphone intravenously in the operating room.
- Fentanyl: Pediatric patients randomized to fentanyl intravenously in the operating room.
Arm/Group | Hydromorphone | Fentanyl
Number analyzed (Participants) | 90 | 90
Participants | 48 | 66

2. Secondary Outcome: Evaluation of Participant's Pain
Description: Revised Face, Legs, Activity, Cry, Consolability (rFLACC) Scale Each of the five categories (F) Face; (L) Legs; (A) Activity; (C) Cry; (C) Consolability is scored from 0-2, which results in a total score between zero and ten. 0=no pain/relaxed, 10=distressed/in pain
Time Frame: Upon arrival and then every 5 minutes for 15 minutes. Then every 15 minutes until discharged from phase 1 of the PACU.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydromorphone | Fentanyl
Number analyzed (Participants) | 90 | 90
score on a scale
  0min | 2.8 (3.5) | 4.3 (3.9)
  5min | 2.7 (3.5) | 3.7 (3.9)
  10min | 2.3 (3.1) | 3.5 (3.6)
  15min | 2.3 (2.5) | 3.4 (3.3)
  30min | 1.7 (2.6) | 2.7 (2.9)
  45min | 0.7 (1.4) | 2.4 (2.4)
  60min | 0.5 (1.1) | 2.1 (2.0)

3. Secondary Outcome: Evaluation of Participant's SpO2 Saturation
Description: SpO2 %
Time Frame: Upon arrival and then every 5 minutes for 15 minutes. Then every 15 minutes until discharged from phase 1 of the PACU.
Measure: Mean (Standard Deviation); unit: percentage of SpO2 saturation
Arm/Group | Hydromorphone | Fentanyl
Number analyzed (Participants) | 90 | 90
percentage of SpO2 saturation
  0min | 96.9 (2.7) | 96.6 (2.7)
  5min | 97.3 (2.8) | 96.1 (9.6)
  10min | 97.4 (2.2) | 97.3 (2.5)
  15min | 97.1 (2.7) | 97.7 (2.1)
  30min | 96.9 (2.1) | 96.8 (9.0)
  45min | 96.8 (2.2) | 97.6 (1.7)
  60min | 96.7 (2.3) | 97.4 (2.0)

4. Secondary Outcome: Respiratory and PONV Events in PACU
Time Frame: up to 6 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Fentanyl
Number analyzed (Participants) | 90 | 90
Participants
  Witnessed apnea in PACU | 3 | 4
  Witnessed desaturation below 90% in PACU | 9 | 11
  PONV in PACU | 1 | 2
  No events | 77 | 73

5. Secondary Outcome: Respiratory and PONV Events at Home
Description: Survey sent to parent by email postoperatively
Time Frame: up to 7 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Fentanyl
Number analyzed (Participants) | 64 | 59
Participants
  Nausea since discharge | 10 | 13
  Vomiting since discharge | 7 | 9
  Problems breathing since discharge | 1 | 2
  No events | 46 | 35

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Hydromorphone; Fentanyl: Pediatric patients will be randomized to receive one of either hydromorphone or fentanyl intravenously in the operating room.
Arm/Group | Hydromorphone | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 15/90 | 12/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone (N=90) | Fentanyl (N=90)
Postoperative tonsillar bleed (Blood and lymphatic system disorders) | 2 | 3 — 5 patients with postoperative tonsillar bleed (2 in the hydromorphone arm, 3 in the fentanyl arm)
Fever (Infections and infestations) | 1 | 1
Prolonged admission for poor oral intake (Gastrointestinal disorders) | 8 | 3
Tongue Injury (Skin and subcutaneous tissue disorders) | 0 | 1
Readmitted for urinary retention (Renal and urinary disorders) | 1 | 0
Readmitted for nausea or vomiting (Gastrointestinal disorders) | 1 | 2
Prolonged admission for nausea or vomiting (Gastrointestinal disorders) | 1 | 2
Postoperative Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04230681/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT04230681/ICF_002.pdf